CLINICAL TRIAL: NCT06877312
Title: Longitudinal Study to Investigate Different Treatment Protocols of Transcranial Electrical Stimulation for Individuals With Dementia
Brief Title: Longitudinal Study to Investigate Different Transcranial Electrical Stimulation
Acronym: tES
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Dr. Zahra Kazem-Moussavi, Professor, Dept. of Electrical and Computer Eng., University of Manitoba
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: B2021:089
Record Dates: First submitted 2025-03-10; First posted 2025-03-14 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-03

CONDITIONS: Dementia; Degenerative, Dementia Mixed
Keywords: dementia, alzheimer, cognitive impairment
MeSH Terms: conditions — Dementia; Mixed Dementias; Cognitive Dysfunction | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (6):
- Transcranial Direct Current Stimulation (tDCS) (Experimental): Participants will receive active tDCS simultaneously with cognitive exercises. It will be optional for participants to have their choice of music playing in the background.
  Interventions: Device: Transcranial Direct Current Stimulation (tDCS)
- 30 Hz Transcranial Alternating Current Stimulation (tACS) (Experimental): Participants will receive active tACS at 30 Hz simultaneously with cognitive exercises. It will be optional for participants to have their choice of music playing in the background.
  Interventions: Device: 30 Hz Transcranial Alternating Current Stimulation (tACS)
- 50 Hz Transcranial Alternating Current Stimulation (tACS) (Experimental): Participants will receive active tACS at 50 Hz simultaneously with cognitive exercises. It will be optional for participants to have their choice of music playing in the background.
  Interventions: Device: 50 Hz Transcranial Alternating Current Stimulation (tACS)
- 70 Hz Transcranial Alternating Current Stimulation (tACS) (Experimental): Participants will receive active tACS at 70 Hz simultaneously with cognitive exercises. It will be optional for participants to have their choice of music playing in the background.
  Interventions: Device: 70 Hz Transcranial Alternating Current Stimulation (tACS)
- 90 Hz Transcranial Alternating Current Stimulation (tACS) (Experimental): Participants will receive active tACS at 90 Hz simultaneously with cognitive exercises. It will be optional for participants to have their choice of music playing in the background.
  Interventions: Device: 90 Hz Transcranial Alternating Current Stimulation (tACS)
- Transcranial Random Noise Stimulation (tRNS) (Experimental): Participants will receive active tRNS simultaneously with cognitive exercises. It will be optional for participants to have their choice of music playing in the background.
  Interventions: Device: Transcranial Random Noise Stimulation (tRNS)

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation (tDCS) — A light electrical current with zero frequency (tDCS) will be applied to the scalp of the participants via 2 electrodes, while the participants perform cognitive exercises with the guidance of a trained research assistant. They have the option of having their choice of music playing in the background while they perform the cognitive exercises.
  Cognitive exercises: Participants will perform memory and learning games/tasks through the "Mind Triggers" app on an IPad and other cognitive games. Participants will be guided by a highly trained research assistant.
  Arms: Transcranial Direct Current Stimulation (tDCS)
Device: 30 Hz Transcranial Alternating Current Stimulation (tACS) — A light electrical current with 30 Hz frequency (tACS) will be applied to the scalp of the participants via 2 electrodes, while the participants perform cognitive exercises with the guidance of a trained research assistant. They have the option of having their choice of music playing in the background while they perform the cognitive exercises.
  Cognitive exercises: Participants will perform memory and learning games/tasks through the "Mind Triggers" app on an IPad and other cognitive games. Participants will be guided by a highly trained research assistant.
  Arms: 30 Hz Transcranial Alternating Current Stimulation (tACS)
Device: 50 Hz Transcranial Alternating Current Stimulation (tACS) — A light electrical current with 50 Hz frequency (tACS) will be applied to the scalp of the participants via 2 electrodes, while the participants perform cognitive exercises with the guidance of a trained research assistant. They have the option of having their choice of music playing in the background while they perform the cognitive exercises.
  Cognitive exercises: Participants will perform memory and learning games/tasks through the "Mind Triggers" app on an IPad and other cognitive games. Participants will be guided by a highly trained research assistant.
  Arms: 50 Hz Transcranial Alternating Current Stimulation (tACS)
Device: 70 Hz Transcranial Alternating Current Stimulation (tACS) — A light electrical current with 70 Hz frequency (tACS) will be applied to the scalp of the participants via 2 electrodes, while the participants perform cognitive exercises with the guidance of a trained research assistant. They have the option of having their choice of music playing in the background while they perform the cognitive exercises.
  Cognitive exercises: Participants will perform memory and learning games/tasks through the "Mind Triggers" app on an IPad and other cognitive games. Participants will be guided by a highly trained research assistant.
  Arms: 70 Hz Transcranial Alternating Current Stimulation (tACS)
Device: 90 Hz Transcranial Alternating Current Stimulation (tACS) — A light electrical current with 90 Hz frequency (tACS) will be applied to the scalp of the participants via 2 electrodes, while the participants perform cognitive exercises with the guidance of a trained research assistant. They have the option of having their choice of music playing in the background while they perform the cognitive exercises.
  Cognitive exercises: Participants will perform memory and learning games/tasks through the "Mind Triggers" app on an IPad and other cognitive games. Participants will be guided by a highly trained research assistant.
  Arms: 90 Hz Transcranial Alternating Current Stimulation (tACS)
Device: Transcranial Random Noise Stimulation (tRNS) — A light electrical current with random noise waveform (tRNS) will be applied to the scalp of the participants via 2 electrodes, while the participants perform cognitive exercises with the guidance of a trained research assistant. They have the option of having their choice of music playing in the background while they perform the cognitive exercises.
  Cognitive exercises: Participants will perform memory and learning games/tasks through "Mind Triggers" app on an IPad and other cognitive games. Participants will be guided by a highly trained research assistant.
  Arms: Transcranial Random Noise Stimulation (tRNS)

SUMMARY:
This research investigates the effect of different frequencies of tACS (0 Hz, 30 Hz, 50 Hz, 70 Hz, 90 Hz) and tRNS with cognitive exercises in a regimen protocol of 4 weeks, everyday (Monday to Friday). The study design is a longitudinal study design in which participants receive different tES randomly ordered. Treatments occur for 4 weeks, then 12 weeks of no treatment (wash-out period), repeated for each tES treatment type. Participants have the option of having their choice of music in the background while they perform cognitive exercises.

DETAILED DESCRIPTION:
This research will investigate the effect of applying transcranial electrical stimulation (tES) with different parameters when paired with cognitive exercises with optional background music on older adults in a longitudinal study. In addition, the researchers will investigate and explore novel technological methods not only to monitor the plausible changes due to intervention. Since most technological interventions on dementia have a demanding and costly protocol, it would be of great interest to personalized optimum treatment strategy. The investigators will use Egocentric Spatial Assessment using our Virtual Reality Navigation (VRN) and functional near infrared spectroscopy (fNIRS) measurements and analysis to develop the monitoring technologies. VRN measures how people orient themselves in a non-familiar environment; the investigators hypothesize that it is deteriorated significantly in Alzheimer's disease even at its onset. fNIRS measures oxygenated and deoxygenated blood flow to the brain and it may help to understand neuronal changes due to intervention.

ELIGIBILITY:
Inclusion Criteria:

* ability to read, write and speak English fluently
* MoCA score between 5 and 24

Exclusion Criteria:

* Being diagnosed with Parkinson's disease, Parkinsonian dementia, Huntington disease, speech significant aphasia and intellectual disability, major depression/anxiety, bipolar disorder, schizophrenia or any other major mood disorder.
* Having a history of epileptic seizures or epilepsy
* Inability to adequately communicate in English
* Impaired vision or hearing severe enough to impair performance in cognitive tests
* Current substance abuse disorder
* Currently participating in another therapeutic study for dementia
* Plan to change the medication during any treatment period (5 weeks including the pre-post assessments)

Ages: 50 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-10-09 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2033-12-31 (Estimated)

PRIMARY OUTCOMES:
Alzheimer's Disease Assessment Scale (ADAS-Cog) | For each tES treatment: Baseline (week 0), Post-treatment (week 5), 1-month follow-up (week 9)
  Change from baseline ADAS-Cog at 5 and 9 weeks. It consists of 11 tasks that include the subject completing tests and observer based assessments. It assesses cognitive domains of memory, language and praxis.
Wechsler Memory Scale (WMS-IV) | For each tES treatment: Baseline (week 0), Post-treatment (week 5), 1-month follow-up (week 9)
  Change from baseline Wechsler Memory Scale (WMS-IV) Older Adult Battery Score at five and nine weeks.
  Cognitive and memory task that focus on 6 major memory indexes: Auditory Memory, Visual Memory, Visual Working Memory, Immediate Memory, Delayed Memory, and Recognition Memory.

SECONDARY OUTCOMES:
N-Back | For each tES treatment: Baseline (week 0), Post-treatment (week 5), 1-month follow-up (week 9)
  N is a number between 1 and 4. A sequence of random shapes is presented and the participant has to tap or say if (remember) whether a presented object is a repeat of the Nth previous object. We will use this test with N=1 as for N>1 is very challenging for dementia population to perform.
Neuropsychiatric Inventory Questionnaire (NPIQ) | For each tES treatment: Baseline (week 0), Post-treatment (week 5), 1-month follow-up (week 9)
  Questionnaire used to assesses neuropsychiatric symptoms and caregiver burden The score of the NPIQ is based on the presence of a specified symptom and a separate score for severity of the symptom. For presence the minimum total score is 0, maximum score is 12. For severity the minimum total score is 0, maximum is 36. Higher scores indicate the participant is exhibiting more severe changes in behaviors.
Functional Near Infrared Spectroscopy (fNIRS) | For each tES treatment: Baseline (week 0), Post-treatment (week 5), 1-month follow-up (week 9)
  fNIRS is a device designed mainly for measuring the blood flow over the prefrontal cortex. Participants will perform a verbal fluency task while the fNIRS measures signals simultaneously.
Virtual Reality Navigation (VRN) spatial orientation test | For each tES treatment: Baseline (week 0), Post-treatment (week 5), 1-month follow-up (week 9)
  The VRN test will be run in non-immersive mode using a large screen and joystick in the PI's office at Riverview Health Center by one of the VRN team member (a research assistant). This program runs only on PC. Run the "rummeego.bat" file in the folder VRN V5 to run the program. Press "s" button to rotate the building. Pressing "Esc" exits that trial and goes to next. The VRN has two stages: 1) Localization, 2) Navigation. The second stage will be carried out only if a participant can pass the localization stage with a score >15 (basically with no consistent side error).

CONTACTS AND LOCATIONS:
Locations (1):
- Riverview Health Centre, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No